CLINICAL TRIAL: NCT05214898
Title: Improving Father-Child and Father-Partner Relationships Through the Evaluation of the 24/7 Dads Intervention With Black and Hispanic Fathers
Brief Title: Improving Father-Child and Father-Partner Relationships Among Black and Hispanic Fathers
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: The Children's Institute (Other); Children's Bureau - Administration for Children and Families (Other)
Responsible Party: Principal Investigator, Julie Cederbaum, Associate Professor, University of Southern California
Other Study IDs: UP-21-00532
Record Dates: First submitted 2021-09-16; First posted 2022-01-31 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Parent-Child Relations; Partner Communication; Parenting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Immediate Start: Investigators will use a quasi-experimental interrupted time series (ITS) design that allows for a continuous sequence of observations on a population, taken repeatedly over time (Bernal et al., 2017). ITS design provides an estimate of the causal effect of a discrete intervention; the design begins with measurements on a dependent variable and the intervention breaks ("interrupts") this time series into preintervention and post-intervention time points. Data will be collected from two group an "Immediate Start Group" and a "Delayed Start Group" (who will serve as a control group for the ITS design).
  Interventions: Behavioral: 24/7 Dad
- Delayed-Start: Investigators will use a quasi-experimental interrupted time series (ITS) design that allows for a continuous sequence of observations on a population, taken repeatedly over time (Bernal et al., 2017). ITS design provides an estimate of the causal effect of a discrete intervention; the design begins with measurements on a dependent variable and the intervention breaks ("interrupts") this time series into preintervention and post-intervention time points. Data will be collected from two group an "Immediate Start Group" and a "Delayed Start Group" (who will serve as a control group for the ITS design).
  Interventions: Behavioral: 24/7 Dad

INTERVENTIONS:
Behavioral: 24/7 Dad — The 24/7 Dad curriculum is an evidence-based, skills driven curriculum (12 group sessions). The following topics are included: Family History, What it Means to Be a Man, Showing and Handling Feelings, Men's Health, Communication, The Father's Role, Discipline, Children's Growth, Getting Involved, Working with & Co-Parenting, Dads and Work, and the "My 24/7Dad Checklist". Healthy Relationship topics include: Communication Skills, including expression, discussion, and negotiation skills; Conflict Resolution and Anger Management; Problem-Solving; and Knowledge of the Benefits of Marriage. Responsible Parenting areas of focus include: children's growth/development; non-violent discipline; co-parenting; building conflict resolutions skills (for the child and the family); and, enhancing family relationships.

SUMMARY:
Fathers play a unique role in the lives of children, with high quality interactions found to improve a child's executive functioning and general school achievement. Father involvement also has positive impacts on fathers themselves, with more involved fathers reporting more self-confidence in their parenting, more satisfaction with parenting, demonstration of more maturity, and reports of less psychosocial distress. However, poverty can have a negative association with fathers parenting and child outcomes, though paternal warmth can mediate this relationship. Children's Institute Inc will recruit and implement the 24/7 Dad program which is designed to provide a comprehensive evidenced-based fatherhood program that builds and strengthens father-child relationships. The curriculum for the primary workshops will be the 24/7 Dad curriculum, which addresses both the responsible parenting and healthy relationship areas in this project. A quasi-experimental interrupted time series (ITS) design allows for a continuous sequence of observations on a population, taken repeatedly over time.

DETAILED DESCRIPTION:
Fathers play a unique role in the lives of children, with high quality interactions found to improve a child's executive functioning and general school achievement. Father involvement also has positive impacts on fathers themselves, with more involved fathers reporting more self-confidence in their parenting, more satisfaction with parenting, demonstration of more maturity, and reports of less psychosocial distress. However, poverty can have a negative association with fathers parenting and child outcomes, though paternal warmth can mediate this relationship. Children's Institute Inc will recruit and implement the 24/7 Dad program which is designed to provide a comprehensive evidenced-based fatherhood program that builds and strengthens father-child relationships. The curriculum for the primary workshops will be the 24/7 Dad curriculum, which addresses both the responsible parenting and healthy relationship areas in this project. The study will use a quasi-experimental interrupted time series (ITS) design that allows for a continuous sequence of observations on a population, taken repeatedly over time. Study aims include: (1) Does the 24/7 Dad intervention influence the behaviors of fathers of young children?; (2) Do fathers who participated in the 24/7 Dad intervention and additional post-intervention support (MIRG and/or financial literacy and job support activities) have better outcomes than those who complete 24/7 Dad only?; (3) Does trauma history and/or current mental wellbeing mediate the relationship between the 24/7 Dad intervention and father engagement, father-child relationships, and co-parenting relationships?; and (4) Does perceived discrimination influence successful outcomes of 24/7 Dad intervention participants? To test the hypotheses of Aim 1 and Aim 2, a generalized linear mixed model will be fitted to the outcome variable individually, specified for corresponding distribution. For Aim 3, investigators will use path models, special cases of structural equation modeling (SEM) with observable variables only, to test the multiple hypothesized mediating pathway.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18 years or older
* Have a child under the age of 24 years
* Speak English or Spanish

Exclusion Criteria:

• Unable to speak English or Spanish

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Program eligibility will be open to all low-income fathers age 18 years or older with children under the age of 24 years. The target geographic area will be South LA, particularly the community of Watts, however participants will not be excluded based on geography. South LA is overwhelmingly Latino (68%) and Black (27%). Close to half (48%) of all residents speak Spanish at home. Nearly all residents are very low-income. We expect our participants to reflect the community in these dimensions.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Father Engagement with Child | 3 months
  Father Engagement Scale (Dyer et al. 2018). 10-item questionnaire measuring interactions between fathers and children

SECONDARY OUTCOMES:
Relationship Conflict | 3 months
  Continuum of Conflict and Control Relationship Scale (Carlson et al., 2017). 20-item scale that identifies variance in relationship IPV, relationship distress, and individual distress
Father-Child Relationship | 3 month
  Child-Parent Relationship Scale - Short Form (Driscoll & Pianta, 2011). 15-item measure of conflict and closeness between fathers and children.
Father Relationship with Co-Parent | 3 months
  Co-Parenting relationship scale (Dyer, Fagan, Kaufman, Pearson, & Cabrera, 2015). 11-item scale aimed at describing the way the father and mother work together as co-parents

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Cederbaum, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
All data will be shared using a unique identifier; no identifying data will be shared